CLINICAL TRIAL: NCT07074171
Title: Addressing COVID-19 Testing Disparities in Vulnerable Populations Using a Community JITAI (Just in Time Adaptive Intervention) Approach: RADx-Underserved Populations (RADxUP) Phase III
Brief Title: Examining How a Text Message-based Educational Intervention Influences COVID-19 Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); University of Texas at Tyler (Other)
Responsible Party: Principal Investigator, Belinda Reininger, Professor and Regional Campus Dean in Brownsville, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-20-1372 Phase 3 Study; U01TR004355 (NIH)
Record Dates: First submitted 2025-07-16; First posted 2025-07-20 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: COVID-19 Testing Behaviors
Keywords: COVID-19; decision making; testing behaviors; vulnerable populations
MeSH Terms: conditions — COVID-19 | interventions — Historically Controlled Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text message-based education intervention (Experimental): A text message-based COVID-19 education intervention with support from community health workers.
  Interventions: Behavioral: Text message-based education intervention
- Historical Control Group (Other): Participants in this Historical Control Group completed the prior Phase II embedded study, in which they received CDC-designed COVID-19 testing brochures and completed pre- and post-intervention surveys only.
  Interventions: Other: Historical Control

INTERVENTIONS:
Behavioral: Text message-based education intervention — The intervention consisted of enhanced behavioral and educational text messages, up to three messages each week, providing updates on COVID-19 testing and vaccination. The text messages included digitally delivered intervention content such as a video with low-literacy instructions for administering the rapid antigen tests, guidance if they tested positive (e.g., quarantine, notify contacts, wearing a mask), and other relevant strategies and content focused on increasing COVID-19 testing and vaccination.
  Arms: Text message-based education intervention
Other: Historical Control — Participants received CDC-designed COVID-19 testing brochures and completed pre- and post-intervention surveys as part of the Phase II embedded study.
  Arms: Historical Control Group

SUMMARY:
In this Phase III study, the investigators will build off of the Phase II embedded study with some adjustments to the design to address new research priorities that examine an intervention that is network informed and delivered through community health worker interactions plus digitally-delivered intervention content with the goal of increasing COVID-19 testing and vaccination. This model, if proven effective, can be scaled up to address COVID-19 and other future pandemics. The investigators will utilize the sample of intervention priority census block groups (PBGs) used in Phase II and will recruit and enroll participants not previously enrolled in either phase I or II from these PBGs using convenience sampling methods. The investigators will use a historical control group consisting of participants from our control arm in Phase II who completed both their baseline and follow-up surveys embedded in the study.

DETAILED DESCRIPTION:
The Phase III study design focuses on vulnerable communities selected to intervention and control conditions and takes advantage of the fact that these communities were randomized to conditions using methods to ensure balanced arms. In Phase III, the investigators will combine the two intervention conditions [Testing Navigation Intervention (TNI) and Facilitated Self-Sampling Intervention (FSSI), and will receive the Multilevel Community network-informed Just-In-Time-Adaptive Intervention (MC-NET-JITAI). The study will include PBGs from each of the two intervention conditions in Phase II; they will be matched to the comparison PBGs on variables such as size, vaccination and testing rates, and the disparities index with the control group. The intervention will last 8 weeks; individuals will be recruited and asked to complete a survey.

Participants who live in a PBG randomized to the intervention arm will be invited to participate in the trial for that arm. In each of the selected intervention PBGs, individuals will be selected via convenience sampling procedures. Recruitment of participants to the MC-NET-JITAI will take place at the participant's home or at one of the community organizations that our participants look to and interact with around COVID-19 topics identified through the social network data. Community Health Workers (CHW) will consent and enroll participants in the MC-NET-JITAI from the randomized PBGs. MC-NET-JITAI will include CHWs providing the participant with a batch of 4 rapid antigen tests that can be shared with people in the household or other close contacts if needed, a COVID-19 resource flier tailored to the study region and updated information about COVID-19 testing and vaccination. The intervention will consist of enhanced behavioral and educational text messages, up to three messages each week, providing updates on COVID-19 testing and vaccination. The text messages will include digitally delivered intervention content such as a video with low-literacy instructions for administering the rapid antigen tests, guidance if they tested positive (e.g., quarantine, notify contacts, wearing a mask), and other relevant strategies and content focused on increasing COVID-19 testing and vaccination. The CHWs will also be available by phone to the participants for any follow-up questions. CHW will follow up via text, email and/or phone with the participants during the two months post-enrollment. In addition to the intervention, the participants will be asked to complete the pre and post-test surveys. Post surveys will be administered online, over the phone, or in person two months after the initial intervention. Study data will be compared to historical control data from the previous phase II Embedded Study.

ELIGIBILITY:
Inclusion Criteria:

* having a smartphone that accepts text messages

Exclusion Criteria:

* having been diagnosed with COVID-19 in the past 30 days based on a positive test (antigen or PCR) or a clinical diagnosis
* having tested for COVID-19 with PCR or antigen test within the past 30 days
* not being available in the recruitment area in the next 60 days
* having been an embedded study participant
* having been a snowball study participant.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Fernandez, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - The University of Texas Health Science Center at Houston School of Public Health Brownsville Regional Campus, Brownsville, Texas
  - The University of Texas Health Science Center at Houston School of Public Health Houston Main Campus, Houston, Texas
  - The University of Texas at Tyler, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Under the protocol, historical controls were not considered enrolled in this study, so they are not included in the enrollment number.
Period: Overall Study
Arm/Group | Text Message-based Education Intervention | Historical Control Group
Started | 384 | 397
Completed | 349 | 397
Not Completed | 35 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text Message-based Education Intervention | Historical Control Group | Total
Number analyzed (Participants) | 384 | 397 | 781
Age, Customized [Count of Participants; unit: Participants]
  <= 18 years | 2 | 4 | 6
  Between 18 and 65 years | 279 | 291 | 570
  >= 65 years | 102 | 91 | 193
  Unknown or Not Reported | 1 | 11 | 12
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 263 | 246 | 509
  Male | 121 | 150 | 271
  Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 259 | 247 | 506
  Not Hispanic or Latino | 125 | 149 | 274
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 384 | 397 | 781

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Self-Reported Use of a COVID-19 Antigen or PCR Test
Description: The number of participants who self-reported use of COVID-19 antigen test or PCR Test using individual-level data in the past 60 days
Time Frame: Baseline
Population: Data were only collected from participants who answered the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Text Message-based Education Intervention | Historical Control Group
Number analyzed (Participants) | 348 | 395
Participants | 31 | 22

2. Primary Outcome: Number of Participants Who Self-Reported Use of a COVID-19 Antigen or PCR Test
Description: as for outcome 1
Time Frame: 8 weeks
Population: Data were only collected from participants who answered the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Text Message-based Education Intervention | Historical Control Group
Number analyzed (Participants) | 348 | 394
Participants | 60 | 46

3. Secondary Outcome: Number of Participants Who Self-reported Receiving COVID-19 Vaccination
Time Frame: Baseline
Population: Data were only collected from participants who answered the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Text Message-based Education Intervention | Historical Control Group
Number analyzed (Participants) | 349 | 395
Participants | 263 | 292

4. Secondary Outcome: Number of Participants Who Self-reported Receiving COVID-19 Vaccination
Time Frame: 8 weeks
Population: Data were only collected from participants who answered the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Text Message-based Education Intervention | Historical Control Group
Number analyzed (Participants) | 349 | 391
Participants | 259 | 12

5. Secondary Outcome: Number of Participants Who Self-reported Used Mitigation Measures if a Positive Test is Obtained
Description: Mitigation measures if a positive test is obtained include mask wearing, isolating, and notifying close contacts.
Time Frame: Baseline, 8 weeks
Population: Data were not collected for this outcome measure because the corresponding question was not included in the study survey. Therefore, no data were available for any participants. This outcome measure will not be collected in the future. The study protocol was not amended to reflect this.
Arm/Group | Text Message-based Education Intervention | Historical Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Text Message-based Education Intervention | Historical Control Group
All-Cause Mortality (participants affected / at risk) | 0/384 | 0/397
Serious Adverse Events (participants affected / at risk) | 0/384 | 0/397
Other Adverse Events (participants affected / at risk) | 0/384 | 0/397

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT07074171/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT07074171/ICF_001.pdf